CLINICAL TRIAL: NCT02153801
Title: Sexual Urinary Function in Patients Undergoing Laparoscopic Low Anterior Resection With Total Mesorectal Excision With High Or Low Ligation of the Inferior Mesenteric Artery With Preservation of Left Colic Artery Multicentre Randomized Trial
Brief Title: Genito Urinary Function With High or Low Inferior Mesenteric Artery Ligation in Laparoscopic Anterior Rectal Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT Number 986
Record Dates: First submitted 2014-05-19; First posted 2014-06-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Genito Urinary Function Evaluation
Keywords: High Ligation, Low ligation, Genito-urinary function, laparoscopy, rectal cancer, aterior resection, Total mesorectal Excision, anastomotic leak.
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Inferior Mesenterci Artery Ligation (Active Comparator): The opening of the peritoneum proceeds cephalad towards the duodenojejunal angle of Treitz, and the mesenteric root is incised 1 cm below the inferior margin of the pancreas. The aortomesenteric window is opened wide and the inferior mesenteric vessels are exposed. The inferior mesenteric artery (IMA) is ligated and divided at 2 cm from its origin. The inferior mesenteric vein is ligated and divided below the pancreatic margin.
  Interventions: Procedure: During the surgical procedure of Laparoscopic Low Anterior Resection with Total mesorectal Excision .
- High Inferior Mesenterci Artery Ligation (Other): For Low Ligation The opening of peritoneum proceeds upward and then laterally towards the sigmoid colon. Left colic artery is identified and preserved while low ligation of the inferior mesenteric artery (superior hemorrhoidal artery) is performed. Lymphadenectomy is carried on medially along the inferior mesenteric artery until 2 cm from the aorta.
  For both groups dissection is then carried on windowing Toldt and Gerota fascias till the parietocolic gutter.
  Interventions: Procedure: During the surgical procedure of Laparoscopic Low Anterior Resection with Total mesorectal Excision .

INTERVENTIONS:
Procedure: During the surgical procedure of Laparoscopic Low Anterior Resection with Total mesorectal Excision . — For High Ligation The opening of the peritoneum proceeds cephalad towards the duodenojejunal angle of Treitz, and the mesenteric root is incised 1 cm below the inferior margin of the pancreas. The aortomesenteric window is opened wide and the inferior mesenteric vessels are exposed. The inferior mesenteric artery (IMA) is ligated and divided at 2 cm from its origin. The inferior mesenteric vein is ligated and divided below the pancreatic margin.
  For Low Ligation The opening of peritoneum proceeds upward and then laterally towards the sigmoid colon. Left colic artery is identified and preserved while low ligation of the inferior mesenteric artery (superior hemorrhoidal artery) is performed. Lymphadenectomy is carried on medially along the inferior mesenteric artery until 2 cm from the aorta.
  For both groups dissection is then carried on windowing Toldt and Gerota fascias till the parietocolic gutter.

SUMMARY:
The aim of this study is to compare the incidence of genito-urinary function depression and anastomotic leak in Laparoscopic Anterior Rectal Resection (LAR) with Total Mesorectal Excision with Ligation if the Inferior Mesenteric Artery at the origin or preserving the Left Colic Artery by a prospective randomized trial.

DETAILED DESCRIPTION:
The level of arterial ligation can affect genito-urinary function (injury to the superior hypogastric plexus), extent (and yield) of lymphadenectomy, distal colonic arterial perfusion (distal colonic arterial perfusion could be deficient due to degenerative disease), sympathic nerve injures. Moreover, colonic stump blood supply together with anastomosis tension are the main factors in developing leaks in rectal surgery and is dependent of the level of ligation. The aim of this study is to compare the incidence of genito-urinary function depression and anastomotic leak in Laparoscopic Anterior Rectal Resection (LAR) with Total Mesorectal Excision with Ligation if the Inferior Mesenteric Artery at the origin or preserving the Left Colic Artery by a prospective randomized trial.

Genito-urinary function will be evaluated with IIEF-5, Internation Consultation Incontinence Modular Questionnarie (ICIQ), Female Sexual Function Index (FSFI), International Index of erectile Function (IIEF) questionnaries and uroflowmetric test pre operatively.

Surgery will be as follow:

The following steps are required in all cases, independently of randomization. The first step consist in the opening of the left part of the gastrocolic ligament and the division of the left part of transverse mesocolon. The splenocolic and phrenocolic attachments are then divided, achieving complete dissection of the left colonic angle. The pelvic peritoneum is opened below the sacral promontory and the hypogastric nerves are identified and preserved. The common iliac veins, the genitofemoral nerve, the gonadic vessels, and the left ureter are successively identified and preserved.

For High Ligation The opening of the peritoneum proceeds cephalad towards the duodenojejunal angle of Treitz, and the mesenteric root is incised 1 cm below the inferior margin of the pancreas. The aortomesenteric window is opened wide and the inferior mesenteric vessels are exposed. The inferior mesenteric artery (IMA) is ligated and divided at 2 cm from its origin. The inferior mesenteric vein is ligated and divided below the pancreatic margin.

For Low Ligation The opening of peritoneum proceeds upward and then laterally towards the sigmoid colon. Left colic artery is identified and preserved while low ligation of the inferior mesenteric artery (superior hemorrhoidal artery) is performed. Lymphadenectomy is carried on medially along the inferior mesenteric artery until 2 cm from the aorta.

For both groups dissection is then carried on windowing Toldt and Gerota fascias till the parietocolic gutter.

Once the descending colonic tract is completely detached from the left parietocolic gutter, dissection of the rectum starts by incision of the peritoneal fold in the pelvis. Total Mesorectal Excision (TME) is then performed according to the principles of Heald.

Colonoscopy will be performed 30 days after surgery to evaluate the anastomosis (leakage, signs of ischemia. Accurate description and pictures of the anastomosis will be produced. IIEF-5, ICIQ, FSFI, International Index of erectile Function (IIEF) and uroflowmetric test will be performed 1 and 9 months post-operatively

ELIGIBILITY:
Inclusion Criteria:

* middle or low rectal cancer (from 0 to 12 cm from the anal verge), American Society Anesthesiologist (ASA) I II III, Body Mass index (BMI) lower than 30.

Exclusion Criteria:

* prior surgery on the abdominal aorta,
* conversion to laparotomy,
* intraoperative decision for colostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Sexual and Urinary Function assessed with with International Prostatic Symptoms Score (IPSS), ICIQ, IIEF, FSFI questionnaires | 9 months from laparoscopic RAR + TME

SECONDARY OUTCOMES:
Incidence of anastomotic leak | 1 month from laparoscopic RAR + TME
Sexual and Urinary Function assessed with with IPSS ICIQ IIEF FSFI questionnaires | 1 month from laparoscopic RAR + TME
Urinary Function assessed with Uroflowmetric examination | 1 months from laparoscopic RAR + TME
Sexual and Urinary Function assessed with with IPSS ICIQ IIEF FSFI questionnaires | 9 month from laparoscopic RAR + TME
Urinary Function assessed with Uroflowmetric examination | 9 months from laparoscopic RAR + TME

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Mari, MD, Study Director
Locations (1):
- Raffaele Pugliese, Milan, Italy

REFERENCES:
- [Derived] Mari GM, Crippa J, Achilli P, Montroni I, Ugolini G, Taffurelli G, Cocozza E, Borroni G, Valenti F, Roscio F, Ferrari G, Origi M, Zuliani W, Pugliese R, Costanzi ATM, Fingherut A, Maggioni D. High Versus Low Ligation of the Inferior Mesenteric Artery During Rectal Resection for Cancer: Oncological Outcomes After Three Years of Follow-Up From the HIGHLOW Trial. Ann Surg Open. 2020 Oct 19;1(2):e017. doi: 10.1097/AS9.0000000000000017. eCollection 2020 Dec. PMID 37637440
- [Derived] Mari G, Santambrogio G, Crippa J, Cirocchi R, Origi M, Achilli P, Ferrari G, Megna S, Desio M, Cocozza E, Maggioni D, Montroni I, Spinelli A, Zuliani W, Costanzi A, Crestale S, Petri R, Bicelli N, Pedrazzani C, Boccolini A, Taffurelli G, Fingerhut A; AIMS Academy Clinical Research Network. 5 year oncological outcomes of the HIGHLOW randomized clinical trial. Eur J Surg Oncol. 2023 Mar;49(3):641-646. doi: 10.1016/j.ejso.2022.10.017. Epub 2022 Oct 28. PMID 36335077
- [Derived] Mari GM, Crippa J, Cocozza E, Berselli M, Livraghi L, Carzaniga P, Valenti F, Roscio F, Ferrari G, Mazzola M, Magistro C, Origi M, Forgione A, Zuliani W, Scandroglio I, Pugliese R, Costanzi ATM, Maggioni D. Low Ligation of Inferior Mesenteric Artery in Laparoscopic Anterior Resection for Rectal Cancer Reduces Genitourinary Dysfunction: Results From a Randomized Controlled Trial (HIGHLOW Trial). Ann Surg. 2019 Jun;269(6):1018-1024. doi: 10.1097/SLA.0000000000002947. PMID 31082897
- [Derived] Mari G, Maggioni D, Costanzi A, Miranda A, Rigamonti L, Crippa J, Magistro C, Di Lernia S, Forgione A, Carnevali P, Nichelatti M, Carzaniga P, Valenti F, Rovagnati M, Berselli M, Cocozza E, Livraghi L, Origi M, Scandroglio I, Roscio F, De Luca A, Ferrari G, Pugliese R. "High or low Inferior Mesenteric Artery ligation in Laparoscopic low Anterior Resection: study protocol for a randomized controlled trial" (HIGHLOW trial). Trials. 2015 Jan 27;16:21. doi: 10.1186/s13063-014-0537-5. PMID 25623323